CLINICAL TRIAL: NCT06299293
Title: Facial Emotion Recognition in Anorexia Nervosa
Acronym: FER_AN
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 21C306
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa
Keywords: Facial emotion recognition; Fear; Anger; Redundant target effect; Alexithymia
MeSH Terms: conditions — Anorexia Nervosa; Affective Symptoms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Participants with Anorexia Nervosa
  Interventions: Other: Facial Emotion Recognition Test
- Controls: Participants with a healthy weight
  Interventions: Other: Facial Emotion Recognition Test

INTERVENTIONS:
Other: Facial Emotion Recognition Test — In this test, the ability to detect and recognize facial expressions of fear or anger will be investigated.

SUMMARY:
Altered emotional processing is reported in Anorexia Nervosa. However, this capability is generally measured through explicit measures, like self-report questionnaires and facial emotion recognition tasks. Instead, no previous research has investigated implicit emotional processing in this clinical condition. In the implicit facial emotion recognition task grounded on the implicit "redundant target effect", individuals generally respond faster when two identical targets are presented simultaneously rather than when presented alone; moreover, the competitive presence of a distractor (that is another emotion or a neutral expression) affects the correct recognition of the target. The ability to recognize and detect facial expressions is explored about two main emotions, fear and anger, because of their role in the intra- and interindividual psychological processing.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* diagnosis of Anorexia Nervosa according to the APA criteria

Exclusion criteria:

- concurrent neurological, neurodevelopmental (e.g., autism), motor, somatosensory and/or psychiatric disorders.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with anorexia nervosa will be recruited at the beginning of a rehabilitative treatment at the Istituto Auxologico Italiano, IRCCS, San Giuseppe Hospital (Italy). Controls will be recruited out of the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Behavioural measure relative to recognition ability | baseline
  Level of accuracy expressed in percentage (min =%; max = 100%) about only the valid trails, in the case of emotion used as target.

SECONDARY OUTCOMES:
Behavioural measure relative to the detection ability | baseline
  Reaction time (i.e., time of response from the onset of the visual stimulus) expressed in milliseconds relative to the valid response for the targeted emotion

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano - Ospedale San Giuseppe, Piancavallo, VCO, Italy